CLINICAL TRIAL: NCT06611761
Title: Prospective Observational Study on the Analgesic Effectiveness of Blocking the Shoulder´s Anterior Capsule and the Suprascapular Nerve by the Anterior Approach Versus Blocking of the Suprascapular and Axillary Nerves by the Posterior Approach in Shoulder Arthroscopy.
Brief Title: Prospective Observational Study on the Analgesic Effectiveness of Blocking the Suprascapular and Axillary Nerves in Shoulder Arthroscopy.
Status: Completed | Type: Observational
Sponsor: Jose Manuel López González (Other)
Responsible Party: Sponsor-Investigator, Jose Manuel López González, Principal investigator, Fundación para la Investigación Biosanitaria del Principado de Asturias
Organization: Fundación para la Investigación Biosanitaria del Principado de Asturias (Other)
Other Study IDs: 2023/491
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Analgesia; Shoulder Arthropathy Associated With Other Conditions; Suprascapular and Axillary Nerve Block
Keywords: shoulder arthroscopy; suprascapular nerve; axillary nerve; multimodal analgesic strategies
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SHAC block + anterior SSN block: Group of patients undergoing shoulder arthroscopy who underwent a block of the anterior capsule of the shoulder (SHAC block) with the suprascapular nerve block (SSN block) performed via an anterior approach with 20 ml of 0.20% ropivacaine
  Interventions: Procedure: Shoulder arthroscopy
- Posterior SSN + AN blocks: Group of patients undergoing shoulder arthroscopy who underwent a suprascapular and axillary nerve block performed via a posterior approach with 20 ml of 0.20% ropivacaine
  Interventions: Procedure: Shoulder arthroscopy

INTERVENTIONS:
Procedure: Shoulder arthroscopy — Shoulder arthroscopy in procedures that cause intense postoperative pain

SUMMARY:
The purpose of this study was to evaluate the analgesic efficacy of suprascapular and axillary nerve block for shoulder arthroscopy surgery

DETAILED DESCRIPTION:
An observational study of paired cohorts, not randomized, was designed with the aim of comparing the postoperative analgesic effectiveness of two regional analgesic techniques: the shoulder anterior capsular block associated with the suprascapular nerve block performed via an anterior approach versus the suprascapular and axillary nerve blocks performed posteriorly in patients with shoulder surgery via arthroscopy in procedures that cause intense postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* ASA (Physical Status Classification System) I - III.
* Having been scheduled for shoulder arthroscopy surgery.

Exclusion Criteria:

Any contraindication for performing regional anesthetic techniques:

* Infection at the puncture point.
* Alteration of hemostasis.
* Allergy to local anesthetics.
* Patient refusal to participate in the study.
* Inability to evaluate postoperative pain.
* Known neuropathy of the operated limb.
* Patients who required conversion to open surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After approval of the study by Galician Drug Research Ethics Committee, Spain (CEIm-G) and obtaining informed consent from the participants, patients undergoing shoulder arthroscopy surgery consecutively over the course of one year were included who met the study inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | The measurement of pain intensity according to the numerical rating scale at preoperative and at the 1st, 2nd, 12th ant 24th postoperative hours
  The measurement of pain intensity according to the numerical rating scale (NRS) from 0 (absence of pain) to 10 (maximum pain endured)

CONTACTS AND LOCATIONS:
Overall Officials: Bárbara María Jiménez Gómez, MD, Principal Investigator — Central University Hospital of Asturias, 33001, Spain
Locations (1):
- FINBA, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Laumonerie P, Dalmas Y, Tibbo ME, Robert S, Faruch M, Chaynes P, Bonnevialle N, Mansat P. Sensory innervation of the human shoulder joint: the three bridges to break. J Shoulder Elbow Surg. 2020 Dec;29(12):e499-e507. doi: 10.1016/j.jse.2020.07.017. Epub 2020 Jul 23. PMID 32712453
- [Background] Yamak Altinpulluk E, Teles AS, Galluccio F, Simon DG, Olea MS, Salazar C, Fajardo Perez M. Pericapsular nerve group block for postoperative shoulder pain: A cadaveric radiological evaluation. J Clin Anesth. 2020 Dec;67:110058. doi: 10.1016/j.jclinane.2020.110058. Epub 2020 Sep 26. No abstract available. PMID 32987232
- [Background] Eckmann MS, Bickelhaupt B, Fehl J, Benfield JA, Curley J, Rahimi O, Nagpal AS. Cadaveric Study of the Articular Branches of the Shoulder Joint. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):564-570. doi: 10.1097/AAP.0000000000000652. PMID 28786899
- [Background] Gonzalez-Arnay E, Jimenez-Sanchez L, Garcia-Simon D, Valdes-Vilches L, Salazar-Zamorano CH, Boada-Pie S, Aguirre JA, Eichenberger U, Fajardo-Perez M. Ultrasonography-guided anterior approach for axillary nerve blockade: An anatomical study. Clin Anat. 2020 May;33(4):488-499. doi: 10.1002/ca.23394. Epub 2019 May 15. PMID 31050830
- [Result] Checcucci G, Allegra A, Bigazzi P, Gianesello L, Ceruso M, Gritti G. A new technique for regional anesthesia for arthroscopic shoulder surgery based on a suprascapular nerve block and an axillary nerve block: an evaluation of the first results. Arthroscopy. 2008 Jun;24(6):689-96. doi: 10.1016/j.arthro.2008.01.019. Epub 2008 Mar 21. PMID 18514113
- [Result] Galluccio F, Fajardo Perez M, Yamak Altinpulluk E, Hou JD, Lin JA. Evaluation of Interfascial Plane and Pericapsular Nerve Blocks to the Shoulder Joint: A Preliminary Analysis of Shoulder Anterior Capsular Block. Pain Ther. 2021 Dec;10(2):1741-1754. doi: 10.1007/s40122-021-00326-0. Epub 2021 Oct 20. PMID 34669181
- [Result] Neuts A, Stessel B, Wouters PF, Dierickx C, Cools W, Ory JP, Dubois J, Jamaer L, Arijs I, Schoorens D. Selective Suprascapular and Axillary Nerve Block Versus Interscalene Plexus Block for Pain Control After Arthroscopic Shoulder Surgery: A Noninferiority Randomized Parallel-Controlled Clinical Trial. Reg Anesth Pain Med. 2018 Oct;43(7):738-744. doi: 10.1097/AAP.0000000000000777. PMID 29659438
- [Result] Sun C, Zhang X, Ji X, Yu P, Cai X, Yang H. Suprascapular nerve block and axillary nerve block versus interscalene nerve block for arthroscopic shoulder surgery: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2021 Nov 5;100(44):e27661. doi: 10.1097/MD.0000000000027661. PMID 34871240

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT06611761/Prot_SAP_ICF_000.pdf